CLINICAL TRIAL: NCT01968603
Title: Weight Gain in Surgically Treated Adult-onset Craniopharyngioma
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zhaoyun Zhang, Clinical Professor, Huashan Hospital
Other Study IDs: KY2013-315
Record Dates: First submitted 2013-10-20; First posted 2013-10-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Adult-onset Craniopharyngioma; Postoperative Weight Gain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study was to describe postoperative weight change in adults undergoing surgery for craniopharyngioma and identify preoperative factors associated with it.

DETAILED DESCRIPTION:
Morbid obesity, intractable weight gain due to hypothalamic damage, is a common and troubling complication in patients undergoing surgery for craniopharyngioma combined or not with radiotherapy, with an incidence of 23~62% in pediatric patients. It has a major negative impact on metabolic and cardiovascular health and quality of life in long-term survivors. Identifying patients at higher risks for developing postoperative weight gain is of great importance in preventing obesity and taking early actions in this population. Though a lot of previous studies have been made in pediatric patients and several factors, such as hypothalamic involvement, higher body mass index (BMI) standard deviation score (SDS) at diagnosis, age at diagnosis and hydrocephalus requiring a shunt, have been identified as risk factors for postoperative weight gain, data on this important morbidity in adult-onset patients are sparse, especially in Chinese population. Therefore, the investigators are going to undertake a retrospective evaluation of postoperative weight change in adult-onset patients undergoing surgery for craniopharyngioma and identify preoperative factors associated with it.

ELIGIBILITY:
Inclusion Criteria:

adult-onset, aged 18 years or more; pathologically confirmed craniopharyngioma; primary surgery performed at our hospital; at least 3 months of follow-up including body weight measurement; ambulatory (since lack of ambulation may predispose to weight gain); not receiving supraphysiologic doses of glucocorticoid (e.g. hydrocortisone, prednisone, or dexamethasone to exceed 12mg/m2•d hydrocortisone equivalent) for more than 2 months after tumor therapy.

Exclusion Criteria:

Childhood-onset, <18 years old; Inconsistent pathology; Without follow-up records in the investigators' institution.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult-onset patients with craniopharyngioma undertaking primary surgery in the investigators' institution
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
percentage of postoperative weight gain | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Li yi ming, Principal Investigator — Huashan Hospital
Locations (1):
- Department of Endocrinology and Metabolism, Shanghai, Shanghai Municipality, China